CLINICAL TRIAL: NCT06101823
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2a Study to Evaluate the Efficacy and Safety of OpSCF in the Treatment of Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Phase 2a Study of Efficacy and Safety of OpSCF in Moderate to Severe Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Opsidio, LLC (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OpSCF-201
Record Dates: First submitted 2023-10-19; First posted 2023-10-26 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Monoclonal Antibody
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OpSCF (Active Comparator): OpSCF, 600 mg, subcutaneously, every two weeks x 14 weeks
  Interventions: Biological: OpSCF
- Placebo (Placebo Comparator): Matched placebo, subcutaneously, every two weeks x 14 weeks
  Interventions: Biological: Placebo
- Open Label Extension (Active Comparator): Subjects may choose to continue in an Open Label Extension (OLE) phase if they complete the randomized phase. All subjects regardless of treatment assignment in the randomized phase will receive OpSCF, 600 mg every 4 weeks for up to 36 weeks.
  Interventions: Biological: OpSCF; Biological: OpSCF (Open Label Extension)

INTERVENTIONS:
Biological: OpSCF — Monoclonal Antibody
  Arms: OpSCF; Open Label Extension
Biological: Placebo — Formulation buffer without active agent
  Arms: Placebo
Biological: OpSCF (Open Label Extension) — Subjects may continue on an Open Label Extension after completing the 16-week randomized portion of the study
  Arms: Open Label Extension

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a monoclonal antibody, OpSCF, in the treatment of adults with moderate to severe Atopic Dermatitis (Eczema). OpSCF will be compared to a placebo.

OpSCF or placebo will be administered every 2 weeks for 14 weeks, and the efficacy will be assessed two weeks later. After that, subjects may choose to enter an Open Label Extension phase in which all subjects will receive OpSCF every 4 weeks for 40 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has clinically confirmed diagnosis of active AD
* Subject has at least a 6-month history of AD
* Subject is willing to use effective birth control

Exclusion Criteria:

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has any clinically significant medical condition that would put the subject at undue risk or interfere with interpretation of study results.
* Subject has used dupilumab within 26 weeks prior to Day 1
* Subject has used tralokinumab within 12 weeks prior to Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percent change in Eczema Area and Severity Index (EASI) score from baseline at Week 16 | 16 weeks
  Validated measure of activity of atopic dermatitis. A score of 0 indicates clear or no eczema, 0.1 to 1.0 indicates almost clear, 1.1 to 7 indicates mild disease, 7.1 to 21 indicates moderate disease, 21.1 to 50 indicates severe disease, and greater than 51 indicates very severe disease.

SECONDARY OUTCOMES:
Incidence of AEs and SAEs | Through study completion, approximately 1 year including the open label extension phase
  Safety
Proportion of subjects achieving at least a 2-grade reduction from baseline to clear (0) or almost clear (1) in vIGA-AD | 16 weeks
  Validated Investigator scoring of AD activity
Change and percent change from baseline in weekly average of the daily Peak Pruritus Numerical Rating Scale (PP-NRS) | 16 weeks
  Validated scale of subject-reported itch. The Peak Pruritus Numerical Rating Scale is a single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours based on the following question: 'On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".

OTHER OUTCOMES:
Change from baseline in blood biomarkers and IgE at Weeks 4, 8, 12, and 16 | 16 weeks
  Blood tests
Change from baseline in skin biomarkers collected using skin biopsies at Weeks 4 and 16 (optional for consenting subjects) | 16 weeks
  Histopathological examination
Change from baseline in skin biomarkers collected using tape strips at Weeks 4 and 16 (optional for consenting subjects) | 16 weeks
  Analysis of proteomics and mRNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Martin Phillips, Study Director — Opsidio, LLC
Locations (22):
- United States (18):
  - Cahaba Dermatology & Skin Health Center, Birmingham, Alabama
  - First OC Dermatology Research, Fountain Valley, California
  - Axon Clinical Research, Inglewood, California
  - University Clinical Trials, San Diego, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Skin Care Research, Boca Raton, Florida
  - Skin Research of South Florida, Miami, Florida
  - RM Medical Research, Miami Lakes, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Options Research Group, West Lafayette, Indiana
  - DS Research of Kentucky, Louisville, Kentucky
  - Oakland Hills Dermatology P.C, Auburn Hills, Michigan
  - Saginaw Bay Dermatology, Bay City, Michigan
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Rodgers Dermatology, Frisco, Texas
  - Dermatology Of Seattle, Bellevue, Washington
- Canada (4):
  - Oshawa Clinic Dermatology Trials, Oshawa, Ontario
  - Research Toronto, Toronto, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No